CLINICAL TRIAL: NCT07198295
Title: Thoracic Endovascular Repair With False Lumen Embolization for Aortic Dissection: A Multicenter, Prospective, Observational Study
Brief Title: TEAVR With False Lumen Embolization for Aortic Dissection
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Hongkun Zhang, MD, Director of the Department of Vascular Surgery, First Affiliated Hospital of Zhejiang University
Other Study IDs: IIT20250894B
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Aortic Dissection Type B
Keywords: Type B aortic dissection; Thoracic endovascular repair; false lumen embolization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: TEVAR with false lumen embolization: Patients with type B aortic dissection who receive TEAVR in the true lumen and vascular plug embolization in the false lumen
  Interventions: Device: TEAVR with false lumen embolization

INTERVENTIONS:
Device: TEAVR with false lumen embolization — The procedure involves two key steps: first, deploying a stent-graft in the true lumen to seal the proximal entry tear; second, selectively catheterizing the false lumen to place 1-3 vascular plugs at critical locations-below the distal end of the stent-graft, at the celiac trunk level, and at the distal re-entry tear in the infrarenal aorta-to occlude distal outflow and induce complete false lumen thrombosis.

SUMMARY:
This multicenter, prospective, observational study aims to evaluate the efficacy and safety of thoracic endovascular aortic repair (TEVAR) combined with false lumen embolization using vascular plugs in patients with acute type B aortic dissection. Despite TEVAR being a standard treatment for type B dissection, long-term outcomes remain suboptimal due to persistent false lumen perfusion through distal re-entry tears, leading to aortic expansion and high reintervention rates. This study addresses the clinical need for a more definitive treatment strategy that promotes complete false lumen thrombosis and aortic remodeling.

The study plans to enroll 72 subjects across multiple centers in China, with each participant followed for 12 months. Key inclusion criteria comprise patients with acute or subacute (≤30 days from onset) type B aortic dissection exhibiting typical symptoms and extending to the infrarenal aorta, who are scheduled for the combined procedure. Exclusion criteria included those requiring emergency surgery, complicated dissections with malperfusion or rupture, trauma-related or infectious etiologies, prior aortic surgery, uncontrolled systemic diseases, recent myocardial infarction or stroke, and patients outside the 18-80 age range or refusing participation.

The primary efficacy endpoint is the complete thrombosis rate of the false lumen in the thoracic aorta at 12 months postoperatively, while the primary safety endpoint is the incidence of major adverse events (MAEs) at the same time point. MAEs are defined as a composite of all-cause mortality, myocardial infarction, respiratory failure requiring prolonged ventilation or reintubation, renal deterioration (>50% reduction in eGFR or new dialysis), bowel ischemia requiring surgery or refractory to medical therapy, major stroke, and grade 3 paraplegia. Secondary endpoints include thrombosis rates at 1 and 6 months in the thoracic aorta, patency and thrombosis status at the celiac trunk and infrarenal aortic levels at 1, 6, and 12 months, incidence of MAEs at earlier timepoints, and rates of endoleaks and reinterventions.

All subjects will receive a standardized treatment protocol involving TEVAR with stent-graft placement to seal the proximal entry tear, followed by selective catheterization of the false lumen and deployment of 1-3 vascular plugs at predetermined locations: one parallel to the distal edge of the thoracic stent-graft, one at the level of the celiac trunk, and one at the distal re-entry tear in the infrarenal aorta. Follow-up assessments are scheduled at 1, 6, and 12 months post-procedure, including clinical evaluation and thoracoabdominal CTA imaging to assess aortic remodeling and complication status.

This investigation represents the first prospective multicenter effort to evaluate the combined TEVAR and false lumen embolization strategy. By addressing the fundamental limitation of conventional TEVAR-incomplete false lumen exclusion-this study may establish a new standard for achieving complete aortic remodeling in type B dissection. The results are anticipated to provide robust evidence for guiding clinical practice and potentially influencing future treatment guidelines in aortic disease management.

ELIGIBILITY:
Inclusion Criteria

Patients must meet all of the following conditions to be enrolled:

1. Diagnosed with acute or subacute (symptom onset ≤30 days) Stanford type B aortic dissection.
2. Present with typical clinical symptoms and imaging-confirmed aortic dissection.
3. Dissection extends distally to involve the infrarenal abdominal aorta.
4. Scheduled to undergo elective TEVAR combined with false lumen embolization.

Exclusion Criteria

Patients will be excluded if they meet any of the following conditions:

1. Requiring emergency surgery due to rupture, impending rupture, or severe malperfusion.
2. Complicated type B dissection (e.g., visceral/limb ischemia, refractory pain, or hemodynamic instability).
3. Suspected traumatic or infectious etiology of the dissection.
4. Previous history of aortic surgery or endovascular repair.
5. Use of alternative techniques during the procedure (e.g., PETTICOAT, long-segment coverage).
6. Uncontrolled systemic diseases (e.g., severe cardiac/pulmonary/hepatic dysfunction, advanced malignancy, cachexia, or uncorrectable coagulation disorders).
7. Myocardial infarction or stroke within the past 6 months.
8. Age <18 years or >80 years.
9. Patient refusal to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll adult patients (aged 18-80 years) diagnosed with acute or subacute uncomplicated type B aortic dissection (TBAD). Participants must exhibit typical clinical and radiological features of TBAD, with distal extension of the dissection to the infrarenal abdominal aorta. All patients are scheduled to undergo elective thoracic endovascular aortic repair (TEVAR) combined with false lumen embolization using vascular plugs.
  The population excludes individuals requiring emergency intervention, those with complicated dissections (e.g., malperfusion, rupture, or refractory pain), previous aortic surgery, trauma- or infection-related etiologies, significant uncontrolled comorbidities, recent major cardiovascular events, or contraindications to the endovascular procedure. The study aims to include a representative sample suitable for evaluating the safety and efficacy of TEAVR with false lumen embolization under real-world clinical conditions.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with complete thrombosis in the false lumen in the thoracic aorta as assessed by CTA | at 12 months postoperatively
Number of participants with major adverse events | at 12 months postoperatively

IPD SHARING:
Plan to Share IPD: No